CLINICAL TRIAL: NCT00106535
Title: A Randomized, Double-blind Study of Safety and Prevention of Structural Joint Damage During Treatment With Tocilizumab Versus Placebo, in Combination With Methotrexate, in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study to Assess the Effect of Tocilizumab + Methotrexate on Prevention of Structural Joint Damage in Patients With Moderate to Severe Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA17823
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Tocilizumab 4 mg/kg + Methotrexate (Experimental): Tocilizumab 4 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly for 52 weeks. From Week 16 participants with < 20% improvement in swollen and tender joints counts were eligible for escape therapy with tocilizumab. After Week 52 participants were able to switch to open label treatment with tocilizumab 8 mg/kg every 4 weeks for 12 months in year 2 (except patients who had a >70% improvement in both swollen and tender joint counts who remained on blinded treatment). Participants who completed year 2 of the study were eligible to enter an optional open-label long-term extension period (Year 3 to 5) and received Tocilizumab 8 mg/kg every 4 weeks.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate
- Tocilizumab 8 mg/kg + Methotrexate (Experimental): Tocilizumab 8 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly for 52 weeks. From Week 16 participants with < 20% improvement in swollen and tender joints counts were eligible for escape therapy with tocilizumab. After Week 52 participants were able to switch to open label treatment with tocilizumab 8 mg/kg every 4 weeks for 12 months in year 2 (except patients who had a >70% improvement in both swollen and tender joint counts who remained on blinded treatment). Participants who completed year 2 of the study were eligible to enter an optional open-label long-term extension period (Year 3 to 5) and received Tocilizumab 8 mg/kg every 4 weeks.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Methotrexate
- Placebo + Methotrexate (Placebo Comparator): Placebo intravenously (IV) every 4 weeks plus methotrexate (MTX) 10-25 mg (oral or parenteral) weekly for 52 weeks. From Week 16 participants with < 20% improvement in swollen and tender joints counts were eligible for escape therapy with tocilizumab. After Week 52 participants were able to switch to open label treatment with tocilizumab 8 mg/kg every 4 weeks for 12 months in year 2 (except patients who had a >70% improvement in both swollen and tender joint counts who remained on blinded treatment). Participants who completed year 2 of the study were eligible to enter an optional open-label long-term extension period (Year 3 to 5) and received Tocilizumab 8 mg/kg every 4 weeks.
  Interventions: Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 4 mg/kg or 8 mg/kg IV/month every 4 weeks.
  Other Names: RoActemra; Actemra
  Arms: Tocilizumab 4 mg/kg + Methotrexate; Tocilizumab 8 mg/kg + Methotrexate
Drug: Placebo — IV/month
  Arms: Placebo + Methotrexate
Drug: Methotrexate — 10-25 mg/week

SUMMARY:
This 3 arm study will compare the safety and efficacy, with respect to a reduction in signs and symptoms and prevention of joint damage, of tocilizumab versus placebo, both in combination with methotrexate (MTX) in patients with moderate to severe active rheumatoid arthritis. Patients will be randomized to receive tocilizumab 4 mg/kg IV, tocilizumab 8 mg/kg IV or placebo IV, every 4 weeks. All patients will also receive methotrexate, 10-25 mg/week. The anticipated time on study treatment is 1-2 years and the target sample size is 500+ individuals. After completion of the 2 year study participants could participate in the optional 3 year open label extension phase (year 3 to 5).

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age with moderate to severe active RA for at least 6 months;
* inadequate response to a stable dose of MTX;
* patients of reproductive potential must be using reliable methods of contraception.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks before entering study, or planned surgery within 6 months after entering study;
* prior treatment failure with an anti-tumor necrosis factor agent;
* women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1196 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (136):
- United States (60):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Santa Maria, California
  - Torrance, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Aventura, Florida
  - Fort Lauderdale, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Idaho Falls, Idaho
  - Meridan, Idaho
  - Chicago, Illinois
  - Rockford, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Frederick, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - St Louis, Missouri
  - Billings, Montana
  - Missoula, Montana
  - Reno, Nevada
  - Dover, New Hampshire
  - Medford, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - Lake Success, New York
  - New York, New York
  - Stony Brook, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Canton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Olympia, Washington
  - Seattle, Washington
  - Glendale, Wisconsin
- Australia (6):
  - Adelaide
  - Malvern
  - Melbourne
  - New Lambton
  - Shenton Park
  - St Leonards
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- China (3):
  - Beijing
  - Nanjing
  - Shanghai
- Denmark (2):
  - Hellerup
  - Odense
- Finland (4):
  - Heinola
  - Helsinki
  - Oulu
  - Vantaa
- France (12):
  - Amiens
  - Bobigny
  - Bois-Guillaume
  - Bordeaux
  - Le Kremlin-Bicêtre
  - Lille
  - Nice
  - Orléans
  - Paris
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
- Greece (2):
  - Athens
  - Heraklion
- Italy (16):
  - Brescia
  - Coppito
  - Florence
  - Genova
  - Milan
  - Napoli
  - Padua
  - Pavia
  - Pisa
  - Reggio Emilia
  - Roma
  - Torino
  - Udine
  - Valeggio sul Mincio
  - Varese
  - Verona
- Mexico (4):
  - Chihuahua City
  - Mexico City
  - Monterrey
  - Obregón
- Norway (3):
  - Haugesund
  - Lillehammer
  - Tromsø
- Poland (9):
  - Bydgoszcz
  - Działdowo
  - Elblag
  - Kalisz
  - Krakow
  - Poznan
  - Szczecin
  - Ustroń
  - Warsaw
- Puerto Rico (2):
  - Ponce
  - San Juan
- South Africa (2):
  - Cape Town
  - Diepkloof
- Spain (6):
  - Barcelona
  - Cadiz
  - Mérida
  - Sabadell
  - Santander
  - Seville
- Switzerland (2):
  - Lausanne
  - Sankt Gallen

REFERENCES:
- [Derived] Khawaja MN, Bergman MJ, Yourish J, Pei J, Reiss W, Keystone E. Routine Assessment of Patient Index Data 3 and the American College of Rheumatology/European League Against Rheumatism Provisional Remission Definitions as Predictors of Radiographic Outcome in a Rheumatoid Arthritis Clinical Trial With Tocilizumab. Arthritis Care Res (Hoboken). 2017 May;69(5):609-615. doi: 10.1002/acr.23008. Epub 2017 Apr 7. PMID 27564431
- [Derived] Kremer JM, Blanco R, Halland AM, Brzosko M, Burgos-Vargas R, Mela CM, Rowell L, Fleischmann RM. Clinical efficacy and safety maintained up to 5 years in patients with rheumatoid arthritis treated with tocilizumab in a randomised trial. Clin Exp Rheumatol. 2016 Jul-Aug;34(4):625-33. Epub 2016 Apr 15. PMID 27087059
- [Derived] Bay-Jensen AC, Platt A, Siebuhr AS, Christiansen C, Byrjalsen I, Karsdal MA. Early changes in blood-based joint tissue destruction biomarkers are predictive of response to tocilizumab in the LITHE study. Arthritis Res Ther. 2016 Jan 20;18:13. doi: 10.1186/s13075-015-0913-x. PMID 26787505
- [Derived] Keystone EC, Anisfeld A, Ogale S, Devenport JN, Curtis JR. Continued benefit of tocilizumab plus disease-modifying antirheumatic drug therapy in patients with rheumatoid arthritis and inadequate clinical responses by week 8 of treatment. J Rheumatol. 2014 Feb;41(2):216-26. doi: 10.3899/jrheum.130489. Epub 2014 Jan 15. PMID 24429164
- [Derived] Siebuhr AS, Bay-Jensen AC, Leeming DJ, Plat A, Byrjalsen I, Christiansen C, van de Heijde D, Karsdal MA. Serological identification of fast progressors of structural damage with rheumatoid arthritis. Arthritis Res Ther. 2013 Aug 14;15(4):R86. doi: 10.1186/ar4266. PMID 23945134
- [Derived] Fleischmann RM, Halland AM, Brzosko M, Burgos-Vargas R, Mela C, Vernon E, Kremer JM. Tocilizumab inhibits structural joint damage and improves physical function in patients with rheumatoid arthritis and inadequate responses to methotrexate: LITHE study 2-year results. J Rheumatol. 2013 Feb;40(2):113-26. doi: 10.3899/jrheum.120447. Epub 2013 Jan 15. PMID 23322466
- [Derived] Wang J, Bansal AT, Martin M, Germer S, Benayed R, Essioux L, Lee JS, Begovich A, Hemmings A, Kenwright A, Taylor KE, Upmanyu R, Cutler P, Harari O, Marchini J, Criswell LA, Platt A. Genome-wide association analysis implicates the involvement of eight loci with response to tocilizumab for the treatment of rheumatoid arthritis. Pharmacogenomics J. 2013 Jun;13(3):235-41. doi: 10.1038/tpj.2012.8. Epub 2012 Apr 10. PMID 22491018
- [Derived] Kremer JM, Blanco R, Brzosko M, Burgos-Vargas R, Halland AM, Vernon E, Ambs P, Fleischmann R. Tocilizumab inhibits structural joint damage in rheumatoid arthritis patients with inadequate responses to methotrexate: results from the double-blind treatment phase of a randomized placebo-controlled trial of tocilizumab safety and prevention of structural joint damage at one year. Arthritis Rheum. 2011 Mar;63(3):609-21. doi: 10.1002/art.30158. PMID 21360490

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was divided into two phases: a 2-year core placebo controlled treatment phase and an optional 3-year extension phase.
Groups:
- Tocilizumab 4 mg/kg + Methotrexate: Tocilizumab (TCZ) 4 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly for 52 weeks. From Week 16 participants with < 20% improvement in swollen and tender joints counts were eligible for escape therapy with tocilizumab. After Week 52 participants were able to switch to open label treatment with tocilizumab 8 mg/kg every 4 weeks for 12 months in year 2 (except patients who had a >70% improvement in both swollen and tender joint counts who remained on blinded treatment). Participants who completed year 2 of the study were eligible to enter an optional open-label long-term extension (LTE) period (Year 3 to 5) and received Tocilizumab 8 mg/kg every 4 weeks.
- All Tocilizumab Exposure + MTX: All tocilizumab (TCZ) exposure + methotrexate (MTX) group included all participants who received at least one dose of tocilizumab during the placebo controlled core study or the long term extension period plus MTX 10-25 mg (oral or parenteral) weekly. Participants received either Placebo, Tocilizumab 4 mg/kg or Tocilizumab 8 mg/kg in the 2 year placebo controlled core treatment phase. In the extension 3 to 5 year period, all participants received 8 mg/kg IV every 4 weeks.
Period: 2-year Placebo Controlled Period
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | All Tocilizumab Exposure + MTX
Started | 394 | 401 | 401 | 0
Intent-to-treat: Received Study Drug | 393 | 399 | 398 | 0
Safety: Actual Treatment Received | 392 | 399 | 399 | 0
Completed Week 24 | 356 | 373 | 366 | 0
Completed Week 52 | 326 | 342 | 338 | 0
Completed | 287 (Completed Week 104 (Year 2). 284 participants randomized to the Placebo arm entered the LTE period.) | 309 (Completed Week 104. 304 participants randomized to the TCZ 4 mg/kg arm entered the LTE period.) | 310 (Completed Week 104. 306 participants randomized to the TCZ 8 mg/kg arm entered the LTE period.) | 0
Not Completed | 107 | 92 | 91 | 0
Period: Long-term Extension Period (Year 3 to 5)
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | All Tocilizumab Exposure + MTX
Started | 0 | 0 | 0 | 894 (Entered the Long-term Extension.)
Completed | 0 | 0 | 0 | 704 (Completed the study.)
Not Completed | 0 | 0 | 0 | 190

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Intent-to-treat population that included all randomized participants who received study drug.
Groups:
- Placebo + Methotrexate: Placebo intravenously (IV) every 4 weeks plus methotrexate (MTX) 10-25 mg (oral or parenteral) weekly.
- Tocilizumab 4 mg/kg + Methotrexate: Tocilizumab 4 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly.
- Tocilizumab 8 mg/kg + Methotrexate: Tocilizumab 8 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly.
- Total: Total of all reporting groups
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate | Total
Number analyzed (Participants) | 393 | 399 | 398 | 1190
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.41) | 51.4 (12.59) | 53.4 (11.72) | 52.0 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 328 | 336 | 325 | 989
  Male | 65 | 63 | 73 | 201

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology-ACR20 Response
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 24
Population: Intent-to-treat (ITT) population included all randomized participants who received study drug. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who received escape therapy, withdrew prematurely or where an ACR could not be calculated, were set to 'Non Responder'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 27.0 | 50.6 | 56.3
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With ACR50 Response
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Week 24
Population: Intent-to-treat population included all randomized participants who received study drug. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who received escape therapy, withdrew prematurely or where an ACR could not be calculated, were set to 'Non Responder'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 9.7 | 25.1 | 32.2
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants With ACR70 Response
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline,Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 2.0 | 11.0 | 12.6
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Swollen Joint Count (66 Joint Count): Mean Change From Baseline at Week 24
Description: 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF was used for swollen joint counts. All assessments were set to missing from the time a patient received escape therapy and only pre-escape therapy joint count assessments were carried forward.
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
joint count
  Baseline Swollen Joint Count (SJC) | 16.6 (9.23) | 17.0 (9.78) | 17.3 (9.48)
  Change from Baseline at Week 24 (n=391,399, 397) | -2.9 (10.37) | -7.9 (9.31) | -9.0 (9.76)

5. Secondary Outcome: Tender Joint Count (68 Joint Count): Mean Change From Baseline at Week 24
Description: 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. LOCF was used for swollen joint counts. All assessments were set to missing from the time a patient received escape therapy and only pre-escape therapy joint count assessments were carried forward.
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
joint count
  Baseline Tender Joint Count (TJC) | 27.9 (14.80) | 27.9 (14.15) | 29.3 (15.22)
  Change from Baseline at Week 24 (n=391,399, 397) | -4.8 (14.61) | -12.2 (14.94) | -14.2 (14.58)

6. Secondary Outcome: Patient's Global Visual Analog Scale (VAS): Mean Change From Baseline at Week 24
Description: The patient's global assessment of disease activity is assessed on a 0 to 100 mm horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. No imputation was used for missing VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
millimeters (mm)
  Baseline Patient Visual Analog Scale (VAS) | 63.1 (23.36) | 61.0 (23.25) | 62.7 (22.49)
  Change from Baseline at Week 24 (n=213,308,316) | -17.5 (26.60) | -25.2 (27.09) | -25.2 (24.95)

7. Secondary Outcome: Physician's Global VAS: Mean Change From Baseline at Week 24
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
mm
  Baseline Physician's Visual Analog Scale (VAS) | 63.1 (17.34) | 62.3 (16.8) | 62.7 (16.90)
  Change from Baseline at Week 24 (n=214,307,320) | -29.0 (24.35) | -36.1 (24.31) | -39.8 (21.82)

8. Secondary Outcome: Patient's Pain VAS: Mean Change From Baseline at Week 24
Description: The patient assessed their pain on a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change indicated improvement.
Time Frame: Baseline and Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. No imputation used for missing VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
mm
  Baseline Patient Pain Visual Analog Scale (VAS) | 55.3 (22.07) | 53.3 (21.97) | 55.7 (22.34)
  Change from Baseline at Week 24 (n=213,308,317) | -12.5 (24.92) | -19.5 (25.24) | -21.8 (25.93)

9. Secondary Outcome: C-Reactive Protein (CRP): Mean Change From Baseline at Week 24
Description: The serum concentration of C-Reactive Protein (CRP) is measured in mg/dL. A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. No imputation was used for missing CRP. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
milligrams/deciliter (mg/dL)
  Baseline C-Reactive Protein (CRP) | 2.235 (2.5068) | 2.076 (2.3892) | 2.337 (2.6065)
  Change from Baseline at Week 24 (n=214,308,321) | -0.3560 (2.12778) | -0.9558 (2.35222) | -2.0699 (2.50035)

10. Secondary Outcome: Erythrocyte Sedimentation Rate: Mean Change From Baseline at Week 24
Description: The Erythrocyte Sedimentation Rate (ESR) was measured in mm/hr. A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. No imputation was used for missing ESR. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: millimeters/hour (mm/hr)
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
millimeters/hour (mm/hr)
  Baseline Erythrocyte Sedimentation Rate (ESR) | 46.5 (24.69) | 45.9 (25.12) | 46.4 (24.8)
  Change from Baseline at Week 24 (n=211,304,318) | -9.5 (24.01) | -21.8 (23.71) | -36.8 (24.12)

11. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI): Mean Change From Baseline at Week 24
Description: HAQ-DI is a self-completed patient questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. Calculate HAQ-DI the patient must have a domain score for at least 6 of 8 domains. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis. No imputation was used for missing HAQ-DI. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Scores on a scale
  Baseline HAQ-DI | 1.5 (0.62) | 1.5 (0.64) | 1.5 (0.60)
  Change from Baseline at Week 24 (n=197,292,301) | -0.32 (0.516) | -0.45 (0.531) | -0.51 (0.580)

12. Primary Outcome: Change From Baseline in Modified Total Sharp-Genant Score at Week 52
Description: Radiographs were taken of each hand and foot at Baseline and Week 52 and evaluated at a central reading service by two independent radiologists using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum total erosion score in the hands is 100 (normalized from 98) and in the feet 42, the maximum scores for joint space narrowing in the hands is 100 (normalized from 104) and in the feet 48. The maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat (ITT) population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Linear extrapolation was used to impute missing week 52 data. Data collected after withdrawal or on escape therapy is excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 290 | 339 | 348
Score on a scale | 1.13 (2.962) | 0.34 (1.451) | 0.29 (1.282)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Van Elteren's test; Stratified by region
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Van Elteren's test; Stratified by region

13. Primary Outcome: Change in Physical Function as Measured by the Area Under the Curve (AUC) for the Change From Baseline in the Health Assessment Questionnaire (HAQ) Disability Index at Week 52
Description: HAQ-DI consisted of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities rated on a 4-point scale where 0=without any difficulty to 3=unable to do. The sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst). Functional disability was determined as a cumulative measure of HAQ-DI over 1 year by using the AUC of the change from baseline in HAQ-DI score through week 52. Decreases in AUC of change from baseline in HAQ-DI indicate a greater average improvement in physical function over time and represent a decrease in sustained impairment. For patients with missing week 52 HAQ-DI score, the AUC of the change from baseline was standardized to 52 weeks using the latest timepoint available for calculation of the AUC. The mean was adjusted for region. A negative change from baseline indicated improvement.
Time Frame: Baseline to Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing HAQ scores. All assessments were set to missing after a patient received escape therapy.
Measure: Least Squares Mean (Full Range); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 366 | 376 | 374
Score on a scale*week | -58.11 (150.839) [-699.8 to 401.0] | -128.37 (165.084) [-1059.6 to 266.8] | -144.06 (173.372) [-895.7 to 323.7]
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for region and original treatment group; Mean Difference (Final Values) = -70.26, 95% CI 2-sided [-96.96 to -43.56]
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for region and original treatment group; Mean Difference (Final Values) = -85.95, 95% CI 2-sided [-112.69 to -59.22]

14. Primary Outcome: Change From Baseline in the Modified Total Sharp-Genant Score at Week 104
Description: Radiographs of each hand and foot were taken at Baseline and Week 104 and evaluated at a central reading service by two independent radiologists using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum total erosion score in the hands is 100 and in the feet 42, the maximum scores for joint space narrowing in the hands is 100 and in the feet 48. The maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Data collected after withdrawal or for patients on escape therapy the data is excluded. Missing data was imputed using linear extrapolation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 1.96 (5.956) | 0.58 (2.357) | 0.37 (1.547)

15. Primary Outcome: Change in Physical Function as Measured by the Area Under the Curve for the Change From Baseline in the Health Assessment Questionnaire- Disability Index (HAQ-DI) at Week 104
Description: HAQ-DI consisted of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities rated on a 4-point scale where 0=without any difficulty to 3=unable to do. The sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst). Functional disability was determined as a cumulative measure of HAQ-DI over 2 years by using the AUC of the change from baseline in HAQ-DI score through week 104. Decreases in AUC of change from baseline in HAQ-DI indicated a gr eater average improvement in physical function over time and represent a decrease in sustained impairment. For patients with missing week 104 HAQ-DI score, the AUC of the change from baseline was standardized to 104 weeks using the latest timepoint available for calculation of the AUC. A negative change from baseline indicated improvement.
Time Frame: Baseline to Week 104
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing HAQ scores. For patients who received escape therapy, the HAQ-DI was set to missing from the time they entered escape.
Measure: Least Squares Mean (Full Range); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 366 | 376 | 374
Score on a scale*week | -139.40 (365.682) [-1503.9 to 801.9] | -287.50 (383.201) [-2145.6 to 630.8] | -320.80 (385.741) [-1776.6 to 677.2]
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for region; Mean Difference (Final Values) = -148.10, 95% CI 2-sided [-205.22 to -90.98]
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for region; Mean Difference (Final Values) = -181.40, 95% CI 2-sided [-238.60 to -124.21]

16. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR20) Response at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 24.7 | 47.9 | 55.8

17. Secondary Outcome: Percentage of Participants With ACR20 Response at Week 104
Description: as for outcome 1
Time Frame: Baseline, Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 29.3 | 49.1 | 54.5

18. Secondary Outcome: Percentage of Participants With ACR50 Response at Week 52
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 10.2 | 30.3 | 36.4

19. Secondary Outcome: Percentage of Participants With ACR50 Response at Week 104
Description: as for outcome 18
Time Frame: Baseline, Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 19.8 | 37.6 | 38.9

20. Secondary Outcome: Percentage of Participants With ACR70 Response at Week 52
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 3.8 | 16.5 | 20.1

21. Secondary Outcome: Percentage of Participants With ACR70 Response at Week 104
Description: ACR50 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 12.2 | 24.3 | 22.4

22. Secondary Outcome: Percentage of Participants With ACR70 Response Maintained for 6 Consecutive Months
Description: as for outcome 20
Time Frame: 104 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 5.6 | 11.5 | 14.3

23. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 52
Description: 66 joints were assessed at Baseline and Week 52 for swelling and joints are classified as swollen/not swollen for a total possible swollen joint count of 0 (best) to 66 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 391 | 399 | 397
Joint count | -2.5 (11.07) | -8.0 (9.95) | -10.2 (10.65)

24. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 52
Description: 68 joints were assessed at Baseline and Week 52 for tenderness and joints were classified as tender/not tender for a total possible tender joint count of 0 (best) to 68 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF was used for missing tender joint data. All assessments were set to missing from the time a patient received escape therapy and only pre-escape therapy joint count assessments were carried forward.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 391 | 399 | 397
Joint count | -4.1 (15.53) | -12.3 (15.74) | -15.6 (16.04)

25. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 52
Description: The patient's global assessment of disease activity is assessed at Baseline and Week 52 using a 0 to 100 mm horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 156 | 248 | 281
Score on a scale | -21.1 (26.22) | -27.2 (28.83) | -29.8 (25.61)

26. Secondary Outcome: Change From Baseline in Physicians Global Assessment of Disease Activity at Week 52
Description: The physician's global assessment of disease activity was assessed using a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing VAS assessments. All assessments were set to missing after the patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 155 | 246 | 279
Score on a scale | -35.2 (25.13) | -42.2 (23.57) | -45.4 (22.22)

27. Secondary Outcome: Change From Baseline in the Patient's Pain VAS at Week 52
Description: The patient assessed their pain at Baseline and Week 52 using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing VAS assessments. Data was set to missing for patients who received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 156 | 248 | 282
Score on a scale | -15.0 (25.10) | -22.9 (25.70) | -26.1 (25.51)

28. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 52
Description: Blood was collected for C-Reactive Protein (CRP) at Baseline and Week 52 and was analyzed at a central laboratory. The serum concentration of CRP was measured in milligrams/deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was made for missing data. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 157 | 247 | 282
mg/dL | -0.3800 (2.50681) | -1.0615 (2.39897) | -2.2584 (2.71950)

29. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 52
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR) at Baseline and Week 52 and was analyzed at a local laboratory. ESR was measured in millimeters/hour (mm/hr). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing data. Data was set to missing for patients who received escape therapy.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 149 | 235 | 274
mm/hr | -10.9 (24.27) | -25.6 (24.68) | -38.5 (24.31)

30. Secondary Outcome: Change From Baseline in Swollen Joint Count at Week 104
Description: 66 joints were assessed at Baseline and Week 104 for swelling and joints were classified as swollen/not swollen for a total possible swollen joint count of 0 (best) to 66 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 391 | 399 | 397
Joint count | -3.5 (11.65) | -9.0 (10.76) | -11.3 (11.31)

31. Secondary Outcome: Change From Baseline in Tender Joint Count at Week 104
Description: 68 joints were assessed for tenderness and joints were classified as tender/not tender for a total possible tender joint count of 0 (best) to 68 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF was used for tender joint counts. All assessments were set to missing from the time a patient received escape therapy and only pre-escape therapy joint count assessments were carried forward.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 391 | 399 | 397
Joint count | -5.9 (17.07) | -13.6 (16.53) | -17.7 (16.73)

32. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 104
Description: The patient's global assessment of disease activity was assessed at Baseline and Week 104 using a 0 to 100 mm horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 137 | 228 | 248
Score on a scale | -33.2 (26.35) | -31.6 (27.05) | -33.9 (26.60)

33. Secondary Outcome: Change From Baseline in Physicians Global Assessment of Disease Activity at Week 104
Description: The physician's global assessment of disease activity was assessed at Baseline and Week 104 using a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 139 | 229 | 250
Score on a scale | -43.9 (21.55) | -49.1 (20.33) | -48.7 (22.20)

34. Secondary Outcome: Change From Baseline in the Patient's Pain VAS at Week 104
Description: The patient assessed their pain at Baseline and Week 104 using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 137 | 228 | 248
Score on a scale | -25.6 (24.44) | -26.6 (25.39) | -28.9 (25.47)

35. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 104
Description: Blood was collected for C-Reactive Protein (CRP) at Baseline and Week 104 and was analyzed at a central laboratory. The serum concentration of CRP was measured in milligrams/deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing data. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 139 | 231 | 251
mg/dL | -1.6346 (2.28001) | -1.6863 (2.20965) | -2.3068 (2.65256)

36. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 104
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR) at Baseline and Week 104 and was analyzed at a local laboratory. ESR was measured in millimeters/hour (mm/hr). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing data. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 139 | 231 | 247
mm/hr | -30.7 (22.26) | -35.4 (25.07) | -36.9 (23.39)

37. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 0.3 Units From Baseline in the HAQ Disability Index at Week 52
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0 (without any difficulty) to 3 (unable to do). HAQ-DI=sum of worst scores in each domain divided by the number of domains answered for a total possible score of 0 (best) to 3 (worst).
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. No imputation was used for missing data. All assessments were set to missing for patients who received escape therapy.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 146 | 235 | 263
Percentage of participants | 52.7 | 59.6 | 62.7

38. Secondary Outcome: Percentage of Participants Who Achieve an Improvement of at Least 0.3 Units From Baseline in the HAQ Disability Index at Week 104
Description: The Stanford Health Assessment Questionnaire disability index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Each domain has at least two component questions. There are four possible responses for each component ranging from 0 (without any difficulty) to 3 (unable to do).HAQ-DI=sum of worst scores in each domain divided by the number of domains answered for a total possible score of 0 (best) to 3 (worst).
  .
Time Frame: Baseline, Week 104
Population: as for outcome 35
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 127 | 218 | 231
Percentage of participants | 58.3 | 63.3 | 62.3

39. Secondary Outcome: Area Under Curve (AUC) of the ACRn to Week 24
Description: The ACRn is defined as each patient's lowest percent improvement from Baseline of 3 measures: tender joint count (68 joints), swollen joint count (66 joints), and the improved score achieved in at least 3 of the 5 remaining ACR core components (physician global assessment, patient global assessment, pain, HAQ, and C-reactive protein or ESR, respectively). AUC of ACRn, a continuous variable, was calculated from Baseline to Week 24. A positive score change from Baseline indicated an improvement. The higher the ACRn score the better.
Time Frame: 24 Weeks
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ score, CRP, ESR and VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 216 | 308 | 320
Score on a scale*week | 609.11 (5551.669) | 2791.49 (5479.514) | 3528.89 (5812.582)

40. Secondary Outcome: Area Under Curve (AUC) of the ACRn to Week 52
Description: The ACRn is defined as each patient's lowest percent improvement from Baseline of 3 measures: tender joint count (68 joints), swollen joint count (66 joints), and the improved score achieved in at least 3 of the 5 remaining ACR core components (physician global assessment, patient global assessment, pain, HAQ, and C-reactive protein or ESR, respectively). AUC of ACRn, a continuous variable, was calculated from Baseline to Week 52. A positive score change from Baseline indicated an improvement. The higher the ACRn score the better.
Time Frame: 52 Weeks
Population: Participants from the Intent-to-treat population(all randomized participants who received study drug) with data available for analysis. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ score, CRP, ESR and VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Least Squares Mean (Full Range); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 156 | 247 | 279
Score on a scale*week | 5551.25 (6080.038) [-49420.8 to 25818.8] | 10763.54 (7488.703) [-74637.5 to 33589.0] | 12644.01 (7248.249) [-13773.8 to 31246.7]
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA; Adjusted for region; Mean Difference (Final Values) = 5212.28, 95% CI 2-sided [3139.40 to 7285.16]
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, ANOVA — Adjusted for region; Mean Difference (Final Values) = 7092.76, 95% CI 2-sided [5066.16 to 9119.36]

41. Secondary Outcome: Area Under Curve (AUC) of the ACRn Score at Week 104
Description: The ACRn is defined as each patient's lowest percent improvement from Baseline of 3 measures: tender joint count (68 joints), swollen joint count (66 joints), and the improved score achieved in at least 3 of the 5 remaining ACR core components (physician global assessment, patient global assessment, pain, HAQ, and C-reactive protein or ESR, respectively). AUC of ACRn, a continuous variable, was calculated from Baseline to Week 104. A positive score change from Baseline indicated an improvement. The higher the ACRn score the better.
Time Frame: 104 Weeks
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 138 | 228 | 249
Score on a scale*week | 21094.97 (22341.489) | 27141.08 (24296.659) | 30876.59 (18177.420)

42. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) at Week 24
Description: The DAS28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity], and ESR. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF was used for tender and swollen joint counts, no imputation used for missing ESR and VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 208 | 301 | 311
Score on a scale | -1.49 (1.257) | -2.45 (1.401) | -3.28 (1.383)

43. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) at Week 52
Description: as for outcome 42
Time Frame: Baseline, Week 52
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 153 | 247 | 273
Score on a scale | -1.88 (1.319) | -2.97 (1.391) | -3.80 (1.263)

44. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) at Week 104
Description: as for outcome 42
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis. LOCF used for tender and swollen joint counts, no imputation used for missing ESR and VAS assessments. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 134 | 223 | 238
Score on a scale | -3.70 (1.416) | -3.82 (1.306) | -4.14 (1.344)

45. Secondary Outcome: Percentage of Participants With DAS28 Good or Moderate EULAR Response at Week 24
Description: The DAS28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] , and ESR. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
  European League Against Rheumatism (EULAR) Good response: DAS28 ≤ 3.2 and a change from Baseline < -1.2.
  EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Baseline, Week 24
Population: ITT population included all randomized participants who received study drug. LOCF was used for tender and swollen joint counts, no imputation used for missing ESR and VAS assessments. For patients who received escape therapy, withdrew prematurely or where the DAS28 score was missing the response was set to 'No response'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants
  Good EULAR Response | 5.9 | 24.6 | 40.7
  Moderate EULAR Response | 28.8 | 39.6 | 33.7

46. Secondary Outcome: Percentage of Participants With DAS28 Good or Moderate EULAR Response at Week 52
Description: The DAS28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm) [visual analog scale: 0=no disease activity to 100=maximum disease activity] , and ESR. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
  European League Against Rheumatism (EULAR) Good response: DAS28 ≤ 3.2 and a change from Baseline < -1.2.
  EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Baseline, Week 52
Population: as for outcome 45
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants
  Good Response | 7.1 | 27.6 | 44.0
  Moderate Response | 22.1 | 30.3 | 24.1

47. Secondary Outcome: Percentage of Participants With DAS28 Good or Moderate EULAR Response at Week 104
Description: as for outcome 46
Time Frame: Baseline, Week 104
Population: ITT population included all randomized participants who received study drug. LOCF was used for tender and swollen joint counts, no imputation was used for missing ESR and VAS assessments. For patients who received escape therapy, withdrew prematurely or where the DAS28 score was missing the response was set to 'No response'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants
  Good Response | 23.4 | 39.6 | 45.7
  Moderate Response | 9.7 | 15.8 | 13.1

48. Secondary Outcome: Percentage of Participants With DAS28 Remission at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR). DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 remission is defined as a DAS28 score <2.6.
Time Frame: Week 24
Population: as for outcome 42
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 212 | 304 | 315
Percentage of participants | 3.8 | 17.8 | 33.3

49. Secondary Outcome: Percentage of Participants With DAS28 Remission at Week 52
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR). DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control.DAS28 Remission is defined as a DAS28 score <2.6.
Time Frame: Week 52
Population: as for outcome 42
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 156 | 249 | 275
Percentage of participants | 7.7 | 30.5 | 48.0

50. Secondary Outcome: Percentage of Participants With DAS28 Remission at Week 104
Description: as for outcome 48
Time Frame: Week 104
Population: as for outcome 42
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 136 | 224 | 241
Percentage of participants | 52.9 | 55.4 | 64.7

51. Secondary Outcome: Area Under Curve (AUC) of Disease Activity Score (DAS28) at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR). DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. Higher calculated AUC values are worse (indicate higher disease activity).
Time Frame: 24 Weeks
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 208 | 301 | 311
Score on a scale*week | 895.85 (179.465) | 767.02 (208.462) | 670.45 (193.506)

52. Secondary Outcome: Area Under Curve (AUC) of Disease Activity Score (DAS28) at Week 52
Description: as for outcome 51
Time Frame: 52 Weeks
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 146 | 230 | 265
Score on a scale*week | 1755.25 (353.653) | 1423.12 (415.188) | 1235.80 (412.134)

53. Secondary Outcome: Area Under Curve (AUC) of Disease Activity Score (DAS28) at Week 104
Description: as for outcome 51
Time Frame: 104 Weeks
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Score on a scale*week
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 134 | 223 | 238
Score on a scale*week | 2793.01 (675.840) | 2426.11 (743.882) | 2094.71 (749.148)

54. Secondary Outcome: Change From Baseline in Modified Total Sharp-Genant Score at Week 24
Description: Radiographs were taken of each hand and foot at Baseline and Week 24 and evaluated at a central reading service by two independent radiologists using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum total erosion score in the hands is 100 and in the feet 42, the maximum scores for joint space narrowing in the hands is 100 and in the feet 48. The maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with Baseline and post-Baseline radiographic data available for this outcome measure. Data collected after withdraw or on escape therapy is excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 283 | 327 | 334
Score on a scale | 0.51 (1.336) | 0.22 (0.843) | 0.19 (0.985)

55. Secondary Outcome: Change From Baseline in Modified Total Sharp-Genant Score at Week 80
Description: Radiographs were taken of each hand and foot at Baseline and Week 80 and evaluated at a central reading service by two independent radiologists using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum total erosion score in the hands is 100 and in the feet 42, the maximum scores for joint space narrowing in the hands is 100 and in the feet 48. The maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 80
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Linear extrapolation was used to impute missing data. Data collected after withdraw or on escape therapy is excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 1.60 (4.658) | 0.46 (1.845) | 0.31 (1.273)

56. Secondary Outcome: Change From Baseline in Erosion Score at Week 24
Description: Radiographs were taken of a total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion for a total possible score of 0 (best) to 142 (worst). A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Data was set to missing for patients who withdrew or received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 283 | 327 | 334
Score on a scale | 0.36 (0.928) | 0.15 (0.563) | 0.11 (0.625)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p = 0.0023, Van Elteren's test; Stratified by region
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Van Elteren's test

57. Secondary Outcome: Change From Baseline in Erosion Score at Week 52
Description: as for outcome 56
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data for this outcome measure. Missing Week 52 data was imputed using Linear extrapolation. Data was set to missing for patients who withdrew or received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 290 | 339 | 348
Score on a scale | 0.71 (1.892) | 0.21 (0.920) | 0.17 (0.860)
Statistical Analysis 1: Comparison: Placebo + Methotrexate vs Tocilizumab 4 mg/kg + Methotrexate; Test type: Superiority or Other; p = 0.0001, Van Elteren's test; Stratified by region
Statistical Analysis 2: Comparison: Placebo + Methotrexate vs Tocilizumab 8 mg/kg + Methotrexate; Test type: Superiority or Other; p < 0.0001, Van Elteren's test; Stratified by region

58. Secondary Outcome: Change From Baseline in Erosion Score at Week 80
Description: as for outcome 56
Time Frame: Baseline, Week 80
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 1.01 (3.101) | 0.27 (1.101) | 0.18 (1.060)

59. Secondary Outcome: Change From Baseline in Erosion Score at Week 104
Description: as for outcome 56
Time Frame: Baseline, Week 104
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 1.24 (3.947) | 0.34 (1.337) | 0.22 (1.301)

60. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score at Week 24
Description: Radiographs were taken of a total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint) for a total possible score of 0 (best) to 148 (worst). A lower change from Baseline indicated a better score.
Time Frame: Baseline, Week 24
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 283 | 327 | 334
Score on a scale | 0.15 (0.659) | 0.07 (0.416) | 0.08 (0.468)

61. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score at Week 52
Description: Radiographs were taken of a total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint) for a total possible score of 0 (best) to 148 (worst). A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Missing data was imputed using linear extrapolation. Data collected after withdraw or on escape therapy was excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 290 | 339 | 348
Score on a scale | 0.42 (1.695) | 0.13 (0.739) | 0.12 (0.640)

62. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score at Week 80
Description: as for outcome 61
Time Frame: Baseline, Week 80
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with Baseline and post-Baseline radiographic data available for this outcome measure. Missing data was imputed using linear extrapolation. Data collected after withdraw or on escape therapy was excluded.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 0.59 (2.589) | 0.19 (1.035) | 0.13 (0.626)

63. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score at Week 104
Description: as for outcome 61
Time Frame: Baseline, Week 104
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Score on a scale | 0.72 (3.321) | 0.24 (1.368) | 0.15 (0.772)

64. Secondary Outcome: Percentage of Participants With no Progression of Erosion at Week 24
Description: Radiographs were taken of a total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion for a total possible score of 0 (best) to 142 (worst). No progression of Erosion score was defined as a change from Baseline of less than or equal to zero.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Data collected after withdraw or on escape therapy was excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 283 | 327 | 334
Percentage of participants | 73.9 | 83.8 | 88.3

65. Secondary Outcome: Percentage of Participants With no Progression of Erosion at Week 52
Description: as for outcome 64
Time Frame: Baseline, Week 52
Population: as for outcome 61
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 290 | 339 | 348
Percentage of participants | 70.0 | 82.6 | 86.8

66. Secondary Outcome: Percentage of Participants With no Progression of Erosion at Week 104
Description: as for outcome 64
Time Frame: Baseline, Week 104
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Missing data was imputed using linear extrapolation. Data collected after withdrawal or on escape therapy was excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Percentage of participants | 71.1 | 78.4 | 85.6

67. Secondary Outcome: Percentage of Participants With no Progression of Joint Space Narrowing at Week 24
Description: Radiographs were taken of a total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint) for a total possible score of 0 (best) to 148 (worst). No progression of Joint Space Narrowing score was defined as a change from Baseline of less than or equal to zero.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline and post-Baseline radiographic data available for this outcome measure. Data collected after withdrawal or on escape therapy was excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 283 | 327 | 334
Percentage of participants | 88.3 | 91.4 | 91.9

68. Secondary Outcome: Percentage of Participants With no Progression of Joint Space Narrowing at Week 52
Description: Radiographs were taken of a total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint) for a total possible score of 0 (best) to 148 (worst). No progression of Joint Space Narrowing score is defined as a change from Baseline of less than or equal to zero.
Time Frame: Baseline, Week 52
Population: as for outcome 66
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 290 | 339 | 348
Percentage of participants | 84.5 | 90.6 | 90.5

69. Secondary Outcome: Percentage of Participants With no Progression of Joint Space Narrowing at Week 104
Description: as for outcome 68
Time Frame: Baseline, Week 104
Population: as for outcome 66
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 294 | 343 | 353
Percentage of participants | 80.3 | 86.0 | 91.2

70. Secondary Outcome: Change From Baseline in HAQ Disability Index (HAQ-DI) at Week 52
Description: HAQ-DI is a self-completed questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. To Calculate HAQ-DI the patient must have a domain score for at least 6 of 8 domains. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing data. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 146 | 235 | 263
Score on a scale | -0.39 (0.570) | -0.52 (0.607) | -0.58 (0.583)

71. Secondary Outcome: Change From Baseline in HAQ Disability Index at Week 104
Description: HAQ-DI is a self-completed questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. To Calculate HAQ-DI the patient must have a domain score for at least 6 of 8 domains. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8). Total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 127 | 218 | 231
Score on a scale | -0.50 (0.612) | -0.58 (0.608) | -0.61 (0.661)

72. Secondary Outcome: Change From Baseline in Quality Life Short Form-36 (SF-36) Score at Week 24
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing data. . Data was set to missing for patients who received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 203 | 283 | 294
Score on a scale
  Physical component score | 5.54 (8.459) | 8.15 (8.135) | 8.46 (8.520)
  Mental component score | 3.27 (11.092) | 4.63 (11.702) | 5.17 (10.869)

73. Secondary Outcome: Change From Baseline in SF-36 Score at Week 52
Description: as for outcome 72
Time Frame: Baseline, Week 52
Population: Participants from the Intent-to-treat population (all participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing data. Data was set to missing for patients who received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 144 | 230 | 261
Score on a scale
  Physical component summary score | 5.6 (8.42) | 9.2 (8.29) | 10.0 (9.13)
  Mental component summary score | 3.7 (10.67) | 5.6 (11.94) | 5.5 (11.49)

74. Secondary Outcome: Change From Baseline in SF-36 Score at Week 104
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 130 | 211 | 228
Score on a scale
  Physical component score | 8.7 (9.53) | 10.1 (9.50) | 9.8 (9.66)
  Mental component score | 5.2 (10.27) | 5.7 (11.22) | 6.2 (11.55)

75. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Score at Week 24
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with data available for analysis. No imputation was used for missing FACIT-Fatigue scores. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 214 | 307 | 313
Score on a scale | 5.32 (10.133) | 7.14 (10.145) | 6.91 (8.877)

76. Secondary Outcome: Change From Baseline in FACIT-F Score at Week 52
Description: as for outcome 75
Time Frame: Baseline, Week 52
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 157 | 250 | 276
Score on a scale | 5.57 (10.087) | 8.14 (10.880) | 8.27 (9.387)

77. Secondary Outcome: Change From Baseline in FACIT-F Score at Week 104
Description: as for outcome 75
Time Frame: Baseline, Week 104
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 138 | 224 | 244
Score on a scale | 6.62 (9.544) | 7.85 (10.578) | 8.63 (9.737)

78. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF) at Week 24 in Those Patients With Positive RF
Description: Blood was collected for Rheumatoid Factor (RF) at Baseline and Week 24 and was analyzed at a central laboratory. RF level was reported in international units/milliliter (IU/mL). A positive RF= >15 IU/mL. A lower number change from Baseline indicated a better result.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) with positive RF at Baseline. No imputation was used for missing data. All assessments were set to missing from the time a patient received escape therapy.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 179 | 252 | 268
IU/mL | -44.7 (273.71) | -79.3 (315.06) | -75.6 (205.76)

79. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF) at Week 52 in Those Patients With Positive RF
Description: Blood was collected for Rheumatoid Factor (RF) at Baseline and Week 52 and was analyzed at a central laboratory. RF level was reported in international units/milliliter (IU/mL). A positive RF= >15 IU/mL. A lower number change from Baseline indicated a better result.
Time Frame: Baseline, Week 52
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 132 | 208 | 232
IU/mL | -21.5 (444.37) | 8.6 (575.02) | -71.6 (213.45)

80. Secondary Outcome: Change From Baseline in Rheumatoid Factor (RF) at Week 104 in Those Patients With Positive RF
Description: Blood was collected for Rheumatoid Factor (RF) at Baseline and Week 104 and was analyzed at a central laboratory. RF level was reported in international units/milliliter (IU/mL). A positive RF= >15 IU/mL. A lower number change from Baseline indicated a better result.
Time Frame: Baseline, Week 104
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 115 | 191 | 206
IU/mL | -29.0 (304.46) | -25.1 (431.29) | -39.2 (253.29)

81. Secondary Outcome: Time to Onset of ACR20 by Treatment Group
Description: Time in days until ACR20 response. ACR20 response was defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: 6 months
Population: Participants from the ITT population [N=393,399,398] (all randomized participants who received study drug) with ACR20 response. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who withdrew, received escape therapy or who did not achieve a response were censored.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 209 | 299 | 328
Days | 116.0 [113.0 to 141.0] | 57.0 [57.0 to 82.0] | 57.0 [56.0 to 57.0]

82. Secondary Outcome: Time to Onset of ACR50 by Treatment Group
Description: Time in days until ACR50 response. ACR50 response was defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: 6 months
Population: Participants from the ITT population [N=393,399,398] (all randomized participants who received study drug) with ACR50 response. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who withdrew, received escape therapy or who did not achieve a response were censored.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 76 | 178 | 205
Days | NA [173.0 to NA] — Value not calculable due to insufficient events. | 170.0 [169.0 to NA] — Value not calculable due to insufficient events. | 141.0 [139.0 to 169.0]

83. Secondary Outcome: Time to Onset of ACR70 by Treatment Group
Description: Time in days until ACR70 response. ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: 6 months
Population: Participants from the ITT population [N=393,399,398] (all randomized participants who received study drug) with ACR70 response. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who withdrew, received escape therapy or who did not achieve a response were censored.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 23 | 89 | 95
Days | NA [NA to NA] — Value not calculable due to insufficient events. | NA [176.0 to NA] — Value not calculable due to insufficient events. | NA [NA to NA] — Value not calculable due to insufficient events.

84. Secondary Outcome: Percentage of Participants Who Withdraw Due to Lack of Sufficient Therapeutic Response
Description: Insufficient therapeutic response (patient not responding to the drug as assessed by the physician) was selected by the investigator as a reason that the patient withdrew from the study.
Time Frame: 104 Weeks
Population: Intent-to-treat population included all randomized participants who received at least 1 dose of study drug. Data on escape therapy is excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 3.1 | 0.3 | 0.5

85. Secondary Outcome: Percentage of Participants in Each Treatment Group Who Receive Escape Therapy
Description: In Escape 1, participants in the Tocilizumab 4 mg/kg + Methotrexate and Tocilizumab 8 mg/kg + Methotrexate groups received tocilizumab 8 mg/kg as escape therapy. Participants in the Placebo + Methotrexate group received tocilizumab 4 mg/kg as escape therapy.
  In Escape 2, all participants received tocilizumab 8 mg/kg.
Time Frame: 104 Weeks
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 392 | 399 | 398
Percentage of participants
  Escape 1 Therapy | 50 | 24 | 15
  Escape 2 Therapy | 8 | 2 | 3

86. Secondary Outcome: Percentage of Participants Who Achieved Remission According to the ACR Remission Criteria by Week 24
Description: The percentage of participants, who achieved ACR remission at any study visit up to Week 24. ACR remission required that all five of the following criteria were met for at least two consecutive months: morning stiffness < 15 minutes, no fatigue, no joint pain, no joint tenderness or pain on motion, no soft tissue swelling in joints or tendon sheaths, and ESR < 30 mm/hr for a female or 20 mm/hr for a male.
Time Frame: 24 Weeks
Population: Intent-to-treat population included all randomized participants who received study drug. LOCF was used for tender and swollen joint counts, no imputation used for morning stiffness, FACIT-Fatigue score, ESR and VAS assessment. Patients with missing data, early withdrawal or who received escape therapy were set to 'Non Responder'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 0.0 | 0.3 | 0.0

87. Secondary Outcome: Percentage of Participants Who Achieved Remission According to the ACR Remission Criteria by Week 52
Description: The percentage of participants, who achieved ACR remission at any study visit up to Week 52. ACR remission required that all five of the following criteria were met for at least two consecutive months: morning stiffness < 15 minutes, no fatigue, no joint pain, no joint tenderness or pain on motion, no soft tissue swelling in joints or tendon sheaths, and ESR < 30 mm/hr for a female or 20 mm/hr for a male.
Time Frame: 52 Weeks
Population: as for outcome 86
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 0.0 | 1.8 | 1.5

88. Secondary Outcome: Percentage of Participants Who Achieved Remission According to the ACR Remission Criteria by Week 104
Description: The percentage of participants who achieved ACR remission at any study visit up to Week 104. ACR remission required that all five of the following criteria were met for at least two consecutive months: morning stiffness < 15 minutes, no fatigue, no joint pain, no joint tenderness or pain on motion, no soft tissue swelling in joints or tendon sheaths, and ESR < 30 mm/hr for a female or 20 mm/hr for a male.
Time Frame: 104 Weeks
Population: as for outcome 86
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 0.0 | 2.0 | 2.5

89. Secondary Outcome: Percentage of Participants Who Achieved Complete Clinical Response at Week 52
Description: Complete clinical response is defined as a continuous 6-month period of remission by ACR criteria [defined as five of the following criteria are met for at least two consecutive months: morning stiffness < 15 minutes, no fatigue, no joint pain, no joint tenderness or swelling, and ESR < 30 mm/hr for a female or 20 mm/hr for a male] and no radiographic progression [defined as change from baseline ≤ 0 in the total Sharp-Genant score, erosion score, and JSN score]. Patients who achieve a complete clinical response at any time in the study are counted as responders, even if the response is not maintained.
Time Frame: 52 Weeks
Population: Intent-to-treat population included all randomized participants who received at least 1 dose of study drug. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments. Patients who received escape therapy, withdrew or where an ACR could not be calculated, were set to 'Non Responder'.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 0.0 | 0.3 | 0.5

90. Secondary Outcome: Percentage of Participants Who Achieved Complete Clinical Response at Week 104
Description: Complete clinical response is defined as a continuous 6-month period of remission by ACR criteria [defined as five of the following criteria are met for at least two consecutive months: morning stiffness < 15 minutes, no fatigue, no joint pain, no joint tenderness or swelling, and ESR < 30 mm/hr for a female or 20 mm/hr for a male] and no radiographic progression [defined as change from baseline ≤ 0 in the total Sharp-Genant score, erosion score, and JSN score].
Time Frame: 104 Weeks
Population: as for outcome 89
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + Methotrexate | Tocilizumab 4 mg/kg + Methotrexate | Tocilizumab 8 mg/kg + Methotrexate
Number analyzed (Participants) | 393 | 399 | 398
Percentage of participants | 0 | 0.3 | 1.0

91. Secondary Outcome: End of Study: Percentage of Participants With ACR Response at Week 260
Description: ACR20/50/70/90 response is defined as a ≥ 20/50/70/90% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant, either C-reactive protein or Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 260
Population: Participants from the Modified Intent-to-treatment population, all exposure group, with data available at Baseline and Week 260. LOCF was used for tender and swollen joint counts, no imputation used for missing HAQ Score, CRP, ESR and VAS assessments.
Measure: Number; unit: Percentage of participants
Groups:
- All Tocilizumab Exposure + MTX: All tocilizumab exposure group included all participants who received at least one dose of tocilizumab during the placebo controlled core study or the long term extension period plus MTX 10-25 mg (oral or parenteral) weekly. Participants received either: placebo, tocilizumab 4 mg/kg or tocilizumab 8 mg/kg in the 2 year placebo controlled core treatment phase. In the extension 3 to 5 year period, all participants received tocilizumab 8 mg/kg IV every 4 weeks.
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 473
Percentage of participants
  ACR 20 Response | 82.9
  ACR 50 Response | 64.9
  ACR 70 Response | 42.1
  ACR 90 Response | 16.7

92. Secondary Outcome: End of Study: Percentage of Participants With DAS28 Remission at Week 260
Description: as for outcome 48
Time Frame: Week 260
Population: Participants from the Modified Intent-to-treatment population, all exposure group, with data available at Week 260. Last observation carried forward was used for tender and swollen joint counts. No imputation used for ESR and Patients Global Assessment of Disease Activity VAS.
Measure: Number; unit: Percentage of participants
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 458
Percentage of participants | 59.4

93. Secondary Outcome: End of Study: Percentage of Participants With DAS28 Low Disease Activity (LDA) at Week 260
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR). DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. LDA is defined as DAS28 ≤3.2.
Time Frame: Week 260
Population: as for outcome 92
Measure: Number; unit: Percentage of participants
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 458
Percentage of participants | 73.8

94. Secondary Outcome: End of Study: Percentage of Participants With DAS28 European League Against Rheumatism (EULAR) Good or Moderate Response at Week 260
Description: The DAS28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28 total scores range from 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement. EULAR Good response: DAS28 ≤ 3.2 and a change from Baseline < -1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Baseline, Week 260
Population: as for outcome 92
Measure: Number; unit: Percentage of participants
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 455
Percentage of participants
  Good Response | 74.1
  Moderate Response | 24.0

95. Secondary Outcome: End of Study: Change From Baseline in Swollen Joint Count at Week 260
Description: 66 joints were assessed at Baseline and Week 260 for swelling and joints are classified as swollen/not swollen for a total possible swollen joint count of 0 (best) to 66 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 260
Population: Participants from the Modified Intent-to-treat population, All Tocilizumab Exposure group, with data available at Baseline and Week 260. Last observation carried forward was used for missing joint counts.
Measure: Mean (Standard Deviation); unit: Joint Count
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 480
Joint Count | -14.2 (10.34)

96. Secondary Outcome: End of Study: Change From Baseline in Tender Joint Count at Week 260
Description: 68 joints were assessed at Baseline and Week 260 for tenderness and joints are classified as tender/not tender for a total possible swollen joint count of 0 (best) to 68 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 260
Population: as for outcome 95
Measure: Mean (Standard Deviation); unit: Joint Count
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 480
Joint Count | -23.6 (14.20)

97. Secondary Outcome: End of Study: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 260
Description: as for outcome 70
Time Frame: Baseline, Week 260
Population: Participants from the Modified Intent-to-treat population, All Tocilizumab Exposure group, with data available at Baseline and Week 260. No imputation was used for missing HAQ score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 444
Score on a scale | -0.58 (0.657)

98. Secondary Outcome: End of Study: Change From Baseline in the Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) at Week 260
Description: as for outcome 32
Time Frame: Baseline, Week 260
Population: Participants from the Modified Intent-to-treat population, all tocilizumab exposure group, with data available at Baseline and Week 260. No imputation was used for missing VAS assessments.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 471
mm | -33.7 (27.22)

99. Secondary Outcome: End of Study: Change From Baseline in the Physician's Global Assessment of Disease Activity VAS at Week 260
Description: as for outcome 26
Time Frame: Baseline, Week 260
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 469
mm | -48.7 (21.70)

100. Secondary Outcome: End of Study: Change From Baseline in the Patient's Pain VAS at Week 260
Description: The patient assessed their pain at Baseline and Week 260 using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 260
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 471
mm | -28.2 (26.78)

101. Secondary Outcome: End of Study: Percentage of Participants With Clinical Improvement in the FACIT-Fatigue Score at Week 260
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a ≥5 change from Baseline.
Time Frame: Baseline, Week 260
Population: Participants from the Modified Intent-to-treat population, All Tocilizumab Exposure group, with data available for analysis at Baseline and Week 260.
Measure: Number; unit: Percentage of participants
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 473
Percentage of participants | 64.1

102. Secondary Outcome: End of Study: Percentage of Participants With Clinical Relevant Improvement in the SF-36 Score at Week 260
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. Clinically relevant improvement is defined as a ≥5 change from Baseline.
Time Frame: Baseline, Week 260
Population: as for outcome 101
Measure: Number; unit: Percentage of participants
Arm/Group | All Tocilizumab Exposure + MTX
Number analyzed (Participants) | 442
Percentage of participants
  Mental Components Summary | 43.7
  Physical Components summary | 69.9

103. Secondary Outcome: End of Study: Change From Baseline in Total Sharp-Genant Score at Week 260
Description: Radiographs were taken of each hand and foot at Baseline and Week 260 and evaluated at a central reading service by two independent radiologists using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint).The maximum total erosion score in the hands is 100 and in the feet 42, the maximum scores for joint space narrowing in the hands is 100 and in the feet 48. The maximum modified Sharp score achievable is 290. A lower number change from Baseline indicated a better score. The results were reported based on the treatment the patient was originally randomized to.
Time Frame: Baseline, Week 260
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline, Week 104 and post-Week 104 radiographic data available for this outcome measure. Linear extrapolation was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Placebo + Methotrexate: Placebo intravenously (IV) every 4 weeks plus methotrexate (MTX) 10-25 mg (oral or parenteral) weekly in the 2 year placebo controlled core treatment phase. In the extension 3 to 5 year period, all participants received tocilizumab 8 mg/kg IV every 4 weeks.
- Tocilizumab + Methotrexate: All participants received at least one dose of tocilizumab during the placebo controlled core study or the long term extension period plus MTX 10-25 mg (oral or parenteral) weekly. Participants received either: placebo, tocilizumab 4 mg/kg or tocilizumab 8 mg/kg in the 2 year placebo controlled core treatment phase. In the extension 3 to 5 year period, all participants received tocilizumab 8 mg/kg IV every 4 weeks.
Arm/Group | Placebo + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 258 | 545
Score on a scale | 3.30 (6.093) | 1.54 (4.272)

104. Secondary Outcome: End of Study: Change From Baseline in Erosion Score at Week 260
Description: Radiographs were taken of a total of 14 locations in each hand and wrist and 6 joints in the foot and were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion for a total possible score of 0 (best ) to 142 (worst). A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Week 260
Population: as for outcome 103
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 258 | 545
Score on a scale | 1.95 (3.640) | 0.83 (2.657)

105. Secondary Outcome: End of Study: Change From Baseline in Joint Space Narrowing Score at Week 260
Description: as for outcome 61
Time Frame: Baseline, Week 260
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with Baseline, Week 104 and post-Week 104 radiographic data available for this outcome measure. Missing data was imputed using linear extrapolation.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 258 | 545
Score on a scale | 1.35 (3.134) | 0.71 (2.222)

ADVERSE EVENTS:
Time Frame: Day 1 thru the End of the Study (Up to 6.0 years).
Description: Safety population included all participants who received study treatment based on the treatment actually received. The number of participants at risk is the number of participants in each arm with an adverse event recorded while receiving that treatment. Participants may be counted in more than one arm.
Groups:
- Placebo + Methotrexate: Placebo intravenously (IV) every 4 weeks plus methotrexate (MTX) 10-25 mg (oral or parenteral) weekly.
  Total Exposure Placebo + MTX = 282.36 patient-years (PY).
- All Tocilizumab 4 mg/kg + Methotrexate: All participants who received tocilizumab (TCZ) 4 mg/kg IV every 4 weeks plus methotrexate (MTX) 10-25 mg (oral or parenteral) weekly during the study.
  Total exposure TCZ 4mg + MTX = 580.99 PY.
- All Tocilizumab 8 mg/kg + Methotrexate: All participants who received tocilizumab 8 mg/kg IV every 4 weeks plus MTX 10-25 mg (oral or parenteral) weekly during the study.
  Total exposure TCZ 8mg + MTX = 3797.94 PY.
Arm/Group | Placebo + Methotrexate | All Tocilizumab 4 mg/kg + Methotrexate | All Tocilizumab 8 mg/kg + Methotrexate
Serious Adverse Events (participants affected / at risk) | 26/392 | 58/599 | 267/1054
Other Adverse Events (participants affected / at risk) | 169/392 | 303/599 | 835/1054
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (N=392) | All Tocilizumab 4 mg/kg + Methotrexate (N=599) | All Tocilizumab 8 mg/kg + Methotrexate (N=1054)
Pneumonia (Infections and infestations) | 2 | 3 | 16
Gastroenteritis (Infections and infestations) | 2 | 2 | 3
Osteomyelitis (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 5
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 7
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 3
Coronary artery disease (Cardiac disorders) | 0 | 1 | 5
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Wegener's granulomatosis (Vascular disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 4
Hypotension (Vascular disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 4
Anaphylactic reaction (Immune system disorders) | 0 | 2 | 1
Transaminases increased (Investigations) | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 10
Bronchitis (Infections and infestations) | 0 | 0 | 5
Diverticulitis (Infections and infestations) | 0 | 0 | 4
Erysipelas (Infections and infestations) | 0 | 0 | 4
Pyelonephritis (Infections and infestations) | 0 | 1 | 3
Appendicitis (Infections and infestations) | 0 | 0 | 3
Arthritis bacterial (Infections and infestations) | 0 | 0 | 3
Bronchopneumonia (Infections and infestations) | 0 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 3
Post procedural infection (Infections and infestations) | 0 | 0 | 3
Septic shock (Infections and infestations) | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 2
Bursitis infective (Infections and infestations) | 0 | 1 | 1
Staphylococcal device related infection (Infections and infestations) | 0 | 0 | 2
Empyema (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 2
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 0
Candida osteomyelitis (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 0 | 1
External ear cellulitis (Infections and infestations) | 0 | 0 | 1
Gallbladder empyema (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1
Mycobacterium chelonae infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1
Prostate infection (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Extranodal marginal zone B-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 8
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 3
Encephalitis (Nervous system disorders) | 0 | 0 | 2
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Demyelination (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Vasculitis cerebral (Nervous system disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 3
Myocardial infarction (Cardiac disorders) | 0 | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 0 | 1
Diffuse vasculitis (Vascular disorders) | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Varicophlebitis (Vascular disorders) | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Bicytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Device dislocation (General disorders) | 0 | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 0 | 4
Chest pain (General disorders) | 0 | 0 | 2
Death (General disorders) | 0 | 0 | 1
Infusion site reaction (General disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Scleroderma renal crisis (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Digital ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palpable purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Corneal perforation (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Methotrexate (N=392) | All Tocilizumab 4 mg/kg + Methotrexate (N=599) | All Tocilizumab 8 mg/kg + Methotrexate (N=1054)
Upper respiratory tract infection (Infections and infestations) | 29 | 55 | 256
Urinary tract infection (Infections and infestations) | 20 | 34 | 170
Nasopharyngitis (Infections and infestations) | 18 | 30 | 123
Hypertension (Vascular disorders) | 12 | 34 | 141
Bronchitis (Infections and infestations) | 21 | 32 | 135
Transaminases increased (Investigations) | 6 | 29 | 97
Influenza (Infections and infestations) | 16 | 19 | 100
Headache (Nervous system disorders) | 8 | 25 | 88
Sinusitis (Infections and infestations) | 10 | 30 | 111
Nausea (Gastrointestinal disorders) | 18 | 19 | 69
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 14 | 105
Diarrhoea (Gastrointestinal disorders) | 10 | 23 | 85
Pharyngitis (Infections and infestations) | 10 | 23 | 103
Alanine aminotransferase increased (Investigations) | 5 | 10 | 66
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 53
Gastroenteritis (Infections and infestations) | 9 | 19 | 82
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 56
Oedema peripheral (General disorders) | 8 | 10 | 64
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 5 | 58
Gastritis (Gastrointestinal disorders) | 5 | 18 | 73
Abdominal pain upper (Gastrointestinal disorders) | 8 | 17 | 53
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 16 | 19 | 99
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 55
Depression (Psychiatric disorders) | 11 | 12 | 60
Contusion (Injury, poisoning and procedural complications) | 6 | 9 | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.